CLINICAL TRIAL: NCT01357447
Title: A Double-blind, Placebo-controlled Cross-over Trial of Pulmozyme for Sjogren's Associated Cough
Brief Title: Pulmozyme for Sjogren's Associated Cough
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No patients enrolled.
Sponsor: UConn Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 11-110-3; 002 (Other: University of CT Health Center)
Record Dates: First submitted 2011-05-18; First posted 2011-05-20 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Sjogren's Syndrome; Cough
Keywords: Sjogren's syndrome; Cough
MeSH Terms: conditions — Sjogren's Syndrome; Cough | interventions — dornase alfa; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dornase alfa (Pulmozyme) (Experimental): Dornase alfa is a highly purified solution of recombinant human deoxyribonuclease I (rhDNase), an enzyme which selectively cleaves DNA.
  Interventions: Drug: Saline
- Saline (Placebo Comparator): Normal saline 0.9% solution
  Interventions: Drug: Dornase alfa; Drug: Saline

INTERVENTIONS:
Drug: Dornase alfa — Dose: 2.5 mg solution BID via nebuliser for 2 weeks
  Other Names: Pulmozyme
  Arms: Saline
Drug: Saline — 2.5 ml via nebuliser BID for 2 weeks (alternating with study drug)

SUMMARY:
Patients with Sjogren's disease have destruction of the mucus secreting cells in the airway. This manifestation of the disease leads to the common complaint of persistent dry cough that is seen in many of these patients. This study is aimed at determining whether the regular use of Pulmozyme will result in decreased cough and improved quality of life.

DETAILED DESCRIPTION:
Patients with Sjogren's disease have destruction of the mucus secreting cells in the bronchi. This manifestation of the disease leads to the common complaint of persistent dry cough that is seen in many of these patients. The investigators theorize that regular use of Pulmozyme will result in decreased cough and improved quality of life, by improving mucus clearance.

Primary Objective:To determine if the use of Pulmozyme, twice a day improves cough-related quality of life or cough severity in patients with chronic cough due to Sjogren's disease.

Secondary Objectives:

1. To determine the DNA content in sputum from patients with chronic cough due to Sjogren's disease.
2. To determine the effect of Pulmozyme use on pulmonary function in patients with chronic cough due to Sjogren's disease.
3. To determine the safety of Pulmozyme, taken twice a day in patients with chronic cough due to Sjogren's disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or above with primary Sjogren's disease (as defined by the American European Consensus Group Criteria), and complaint of chronic cough.
* Able to give consent and anticipated ability to adhere to the study procedures.

Exclusion Criteria:

* Diagnosis of COPD, emphysema, asthma, chronic bronchitis, other clinically significant lung disease that is likely to cause cough. Interstitial lung disease associated with Sjogren's is not excluded.
* Cigarette use of greater than 20 pack years or regular use within 6 months
* Allergy or intolerance to Pulmozyme.
* Acute respiratory infection or other acute respiratory illness during the prior month.
* LCQ greater than 17 and VAS less than 3 cm at baseline (Visit 1).
* Pregnancy or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-05; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Changes in Leicester Cough Questionnaire (LCQ) score and cough visual analog scale. | After 2 weeks of therapy.
  To determine if the use of Pulmozyme, twice a day improves cough-related quality of life or cough severity in patients with chronic cough due to Sjogren's disease.

SECONDARY OUTCOMES:
Change in spirometry, specifically FEV1, FVC, FEV1/FVC and FEF 25-75% | After 2 weeeks of therapy
  Changes in pulmonary function in study subjects with use of pulmozyme will be determined by measuring specific spirometric indices (FEV1, FVC, FEV1/FVC and FEF 25-75%)
To determine the DNA content in sputum from patients with chronic cough due to Sjogren's disease. | At start of study
  Sputum from patients with chronic cough due to Sjogren's disease will be analyzed to determine the DNA content at the start of the study.
To determine the safety of Pulmozyme, taken twice a day in patients with chronic cough due to Sjogren's disease. | After 2 weeks of therapy.
  Adverse reactions, if any, due to use of Pulmozyme, taken twice a day in study patients, will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Metersky L Mark, MD, Principal Investigator — University of CT Health Center
Locations (1):
- University of CT Health Center, Farmington, Connecticut, United States